# Document: Protocol and Statistical Analysis Plan

Official Study Title: Prostate Cancer – Comparative Outcomes of New Conceptual Paradigms for Treatment

NCT #: 04890314

IRB Protocol #: 20-08022531

Document Date: Sep 13, 2021

TITLE: Prostate Cancer Comparative Outcomes of New Conceptual Paradigms for

Treatment

IRB Protocol #: 20-08022531

Version Date: 13Sep2021

Funding Source: Patient-Centered Outcomes Research Institute (PCORI)

Principal Investigator: Jim C. Hu, MD MPH

Weill Cornell Medicine

525 E. 68th Street, Starr 946

New York, NY 10065 Phone: 646-962-9600 Fax: 646-962-0715

<u>Jch9011@med.cornell.edu</u>

Ronald C. Chen, MD MPH

University of Kansas

4001 Rainbow Blvd, MS 4033

Kansas City, KS 66160 Phone: 913-588-3612 <u>Rchen2@kumc.edu</u>

Co-Investigators: Ann S. Hamilton, PhD

University of Southern California

2001 N. Soto Street, SSB 318E

Los Angeles, CA 90033 Phone: 323-865-0434 ahamilt@med.usc.edu

Maria Schymura, PhD

New York State Department of Health

150 Broadway, Suite 361

Albany, NY 11204 Phone: 518-474-2255

Maria.schymura@health.ny.gov

Statistician: Andrew J. Vickers, PhD

Memorial Sloan Kettering Cancer Center

485 Lexington Ave, 2<sup>nd</sup> Floor

New York, NY 10017 Phone: 646-888-8233 vickersa@mskcc.org

## **Table of Contents**

| List of Abbreviations | iv |
|-------------------------------------------------------------------------|----|
| 1. Protocol Summary | 1 |
| 1. Study Objectives | |
| 1.1. Objectives | |
| 1.2 Hypotheses / Research Questions | 2 |
| 2. Background and Significance | 3 |
| 3. Study Design and Methods | 3 |
| 3.1 Overall Design | 3 |
| 3.2 Patient Questionnaires – Refer to Appendix A | 3 |
| 4. Study Enrollment | 4 |
| 4.1 Study Population | 4 |
| 4.2 Inclusion Criteria | 4 |
| 4.3 Exclusion Criteria | 4 |
| 4.4 Recruitment and Retention | 4 |
| 6. Study Procedures | 5 |
| 6.1 Schedule of Trial Events | 5 |
| 7. Data Reporting / Regulatory Considerations | 5 |
| 7.1 Institutional Review Board/Ethics Committee Approval | 6 |
| 7.2. Ethical Conduct of the Study | |
| 7.3 Informed Consent | |
| 7.4 Compliance with Trial Registration and Results Posting Requirements | |
| 8. Statistical Considerations | 7 |
| APPENDIX A | 9 |
| Baseline Survey | C |
| First Follow Up Survey | |
| Second Follow Un Survey | |

| Confiden | tiality | Statem | ent |
|----------|---------|--------|-----|
|----------|---------|--------|-----|

| | is to be distributed for review only to in | • . |
|---|---|---|
| | taff, and applicable independent ethics<br>ontents of this document shall not be dis | |
| written authorization from WCM. | | |
| Institution Name | | |
| Principal Investigator's Name | Principal Investigator's Signature | Date |

#### **List of Abbreviations**

AE Adverse Event
AS Active surveillance
BMI Body Mass Index

**CER** Comparative Effectiveness Research

**CFR** Code of Federal Regulations

CI Confidence interval CRF Case Report Form

CTSC Clinical Translational Science Center

**FDA** Food and Drug Administration

**GCP** Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act of 1996

**HRQOL** Health Related Quality of Life

ICF Informed Consent Form

IMRT Intensity Modulated Radiation Therapy

IRB Institutional Review Board

NCCN National Comprehensive Cancer Network

NYS New York State

PCORI Patient-Centered Outcomes Research Institute

PC-CONCEPT Prostate Cancer Comparative Outcomes of New Conceptual

Paradigms for Treatment

**PGA** Partial Gland Ablation

PHI Protected Health Information

PI Principal Investigator
PSA Prostate-specific antigen

**REDCap** Research Electronic Data Capture

RP Radical Prostatectomy
SAC Study Advisory Committee

SBRT Stereotactic Body Radiation Therapy

SCa Southern California

**SEER** Surveillance Epidemiology and End Results

WCM Weill Cornell Medicine

#### 1. Protocol Summary

Full Title: Prostate Cancer Comparative Outcomes of New Conceptual

Paradigms for Treatment

Short Title: PC CONCEPT

Principal Investigators: Jim C. Hu, MD MPH; Ronald C. Chen, MD MPH

**Study Description:** This study will use a population-based cohort design to study men

with newly diagnosed low- and intermediate-risk prostate cancer at high-volume centers in Southern California (SCa) and New York State (NYS). Complications of contemporary treatments for prostate cancer and quality of life outcomes, such as general health, urinary, sexual, and bowel function, cancer anxiety, and treatment regret will be compared and tracked over the course of

this study.

Sample Size: N= 3,657

**Enrollment:** This study will enroll 2,378 subjects and screen up to 3,657

subjects.

Study Population: Subjects will have pathologically-confirmed clinically localized

prostate adenocarcinoma with National Comprehensive Cancer Network (NCCN) low (T1-T2a, Gleason 6, Grade Group 1, PSA <10 ng/mL) or intermediate risk (T2b-T2c or, Gleason 7, Grade Group 2 or 3 or PSA 10-20 ng/mL) at one of the selected hospitals in SCa and NYS. Subjects must also have a diagnosis date during

the 18-month recruitment window.

**Enrollment Period:** 18 months

**Study Design:** Prospective, observational

**Description of Sites** Patient enrollment at 15 sites within SCa and NYS, identified

through National Cancer Institute-sponsored Surveillance

Epidemiology and End Results (SEER)

**Study Duration:** 01Oct2020 - 30Nov2023

Participant Duration: 12 months

**Primary Objectives:** To measure the self-reported, overall and disease specific health

related quality of life (HRQOL) prior to treatment, at 8 months, and 12 months following active surveillance (AS), SBRT, IMRT, PGA,

and RP.

To define and compare the rate of adverse events following stereotactic body radiation therapy (SBRT), partial gland ablation (PGA), intensity modulated radiation therapy (IMRT) and radical prostatectomy (RP) among men recently diagnosed with low and intermediate risk prostate cancer.

#### **Primary Endpoints:**

Change from Baseline in Patient-Reported Quality of Life as Measured on EQ-5D-5L at 8 Months & 12 Months following Treatment

Change from Baseline in Patient-Reported Urinary, Sexual, and Bowel Function as Measured on EPIC-26 at 8 Months & 12 Months following Treatment

Change from Baseline in Ejaculatory Function as Measured on MSHQ-EjD at 8 Months & 12 Months following Treatment

Change from Baseline in Patient-Reported Anxiety as Measured on MAX-PC at 8 Months & 12 Months following Treatment

Assessment of Treatment Regret as Measured on Clark's Prostate Cancer Health Worry at 8 Months & 12 Months following Treatment

Assessment of Adverse Events at 8 Months & 12 Months following Treatment by CTCAE v5.0

Assessment of Cancer Recurrence at 8 Months & 12 Months following Treatment by Patient Medical Records

#### 1. Study Objectives

To compare complications of contemporary treatments for prostate cancer and quality of life outcomes in men with newly diagnosed low- and intermediate-risk prostate cancer through a prospective, population-based cohort study design.

#### 1.1. Objectives

To measure the self-reported, overall and disease specific health related quality of life (HRQOL) prior to treatment, at 8 months, and 12 months following active surveillance (AS), SBRT, IMRT, PGA, and RP.

To define and compare the rate of adverse events following stereotactic body radiation therapy (SBRT), partial gland ablation (PGA), intensity modulated radiation therapy (IMRT) and radical prostatectomy (RP) among men recently diagnosed with low and intermediate risk prostate cancer.

#### 1.2 Hypotheses / Research Questions

PGA is associated with less reduction of urinary and sexual function compared to before treatment than both RP and IMRT. SBRT is associated with less reduction of urinary and sexual

function before treatment compared to RP and IMRT. SBRT will be associated with less reduction in bowel function compared to IMRT. PGA is associated with better overall quality of life at 12 months compared to AS.

PGA and SBRT are associated with fewer adverse events compared to RP and IMRT.

#### 2. Background and Significance

Prostate cancer remains the most commonly diagnosed, solid organ tumor and the second most common cause of cancer death in U.S. men. Technological advances have enabled new treatment options, such as stereotactic body radiation therapy (SBRT) and partial gland ablation (PGA). Although heavily marketed as more convenient with fewer side effects, there is an absence of high-level, comparative effective research (CER) to discern relative outcomes to traditional therapies such as active surveillance (AS), radical prostatectomy (RP) and intensity modulated radiation therapy (IMRT).

We will conduct a pragmatic, population-based cohort study of men with newly diagnosed low and intermediate risk prostate cancer in Southern California (SCa) and New York State (NYS) Surveillance Epidemiology and End Results (SEER) regions to bridge the evidence gap concerning adverse events and patient reported outcomes. Our proposed study will inform multiple stakeholders, who contributed to our study design. This includes prostate cancer survivors, payers, medical device manufacturers, professional organizations, community and academic prostate cancer experts and the Food and Drug Administration (FDA).

#### 3. Study Design and Methods

#### 3.1 Overall Design

We will conduct rapid case ascertainment (within 3 weeks of diagnosis or sooner) at hospitals within these National Cancer Institute-sponsored Surveillance Epidemiology and End Results (SEER) Regions where PGA and SBRT are more likely to be offered. Cases will be identified through the SEER registries' rapid case ascertainment system, and patients will be enrolled to the cohort study directly by the investigator team (not through the individual hospitals). At the time of rapid case ascertainment, the type of treatment a man receives is not yet known; therefore, we will enroll all patients diagnosed with low and intermediate-risk prostate cancer.

### 3.2 Patient Questionnaires - Refer to Appendix A.

#### A. Administration

 Timing and Frequency – Baseline questionnaires will be sent to eligible participants for study enrollment. Follow-up questionnaires at 8 months and 12 months will be sent to enrolled participants to ascertain treatment choice and obtain patient-reported outcomes following treatment.

#### Survey method

Eligible participants will be mailed a survey packet consisting of a paper copy of the survey, an introductory letter and information sheet, and a postage paid return envelope. In the letter the participant will be informed that, if he wishes, he may also complete the survey online and will be given a code and link to the online survey. All materials will be provided in Spanish and English to those participants with Spanish surnames. Interviewers contacting the men are bilingual.

A modified Dillman method will be used to increase response. This includes follow-up with telephone, mail, and offers of completion of the survey online or by telephone.

Specifically, if no response is received after 2 weeks, the study staff will telephone the participant to determine if he has any questions or concerns and to encourage him to complete the survey. At least 5 calls will be made on different days, times of the day (including evenings), and on weekends to reach the person. Additional follow-up efforts will include sending reminder postcards, re-mailing of the survey packet, sending a reminder letter with the link to the online survey, or offering to do the interview over the telephone.

#### Person Identifiers

Patient identifiers obtained at the time of rapid case ascertainment will be used to link to the completed registry abstract. The registry variables to be linked to the cases will include: patient demographic data (age, date of birth, race, socio-economic status, quintile of census block of residence, marital status, birthplace), tumor data (PSA, stage, histology, grade, clinical and pathologic Gleason score, extension), treatment data (surgical code, radiation (type), dates of treatments, chemotherapy, and hormone therapy, PGA and AS).

#### B. Study Instruments – Refer to **Appendix A.**

#### 4. Study Enrollment

#### 4.1 Study Population

Subjects with a diagnosis of prostate cancer who meet the inclusion and exclusion criteria will be eligible for participation in this study.

#### 4.2 Inclusion Criteria

To be included in the study, the participant will: (1) have pathologically-confirmed clinically localized prostate adenocarcinoma with Grade Group 1-2 (Gleason score 6 & 7)<sup>72</sup> at one of the selected hospitals in SCa and NYS; (2) have a diagnosis date during the 18 month recruitment window; (3) speak either English or Spanish and; 4) agree to participate by completing the baseline questionnaire.

#### 4.3 Exclusion Criteria

Patients will be **excluded** if they: 1) have clinically metastatic disease or high-risk PCa (T3a-T4, Gleason Grade Group 4 or 5 or PSA >20 ng/mL; (2) do not speak English or Spanish; or (3) are unwilling or unable (low literacy, too ill, etc.) to give informed consent; or (4) are diagnosed with prostate cancer incidentally at the time of radical cysto-prostatectomy to treat bladder cancer.

#### 4.4 Recruitment and Retention

We will conduct rapid case ascertainment (within usually 4 weeks of diagnosis or sooner) at hospitals within these SEER Regions where PGA and SBRT are more likely to be offered in order to maximize the sample size of men receiving these new treatments.

The SCa and NYS SEER registries are mandated by their respective states to routinely collect and report information on all cancers diagnosed in their catchment areas, including sociodemographic information and tumor characteristics, such as final pathologic stage and histologic grade. Active and passive follow-up is also conducted to ascertain vital status and underlying cause of death.

The Study Advisory Committee (SAC) is comprised of patient partners Fans for the Cure and Us TOO, a senior FDA officer, and a representative from Centers for Medicare and Medicaid Services. Patient partners will participate actively in research decision-making through monthly SAC meetings. Patient partners will co-lead to troubleshoot challenges that may arise in subject recruitment, review preliminary outcomes, troubleshoot research obstacles and participate in dissemination of study findings. Patient partners will resolve potentially confusing and/or missing survey responses.

#### 6. Study Procedures

| 6.1 Sc | hedule | of Trial | l Events |
|--------|--------|----------|----------|
|--------|--------|----------|----------|

| Data elements | Baseline | 8<br>months | 12<br>months |
|-------------------------------------|----------|-------------|--------------|
| Patient reported | | | |
| Income | Χ | | |
| Education | X | | |
| Family history of prostate cancer | Χ | | |
| Employment status | Χ | X | Χ |
| Charlson co-morbidity | Χ | X | X |
| Height | Χ | X | X |
| Weight | X | X | Χ |
| Medications | X | X | X |
| Treatment (confirm PGA and SBRT) | | | |
| Cancer recurrence | | X | X |
| Secondary treatment(s) | | X | Χ |
| Adverse events | | X | Χ |
| Patient reported outcomes | Χ | X | X |
| Registry reported | | | |
| Age | Χ | | |
| Race | Χ | | |
| Marital status | Χ | | |
| Insurance type | X | | |
| Poverty level based on census tract | X | | |
| PSA | Χ | | |
| Biopsy pathology | X | | |
| Clinical stage | Χ | | |
| Treatment | Χ | | |

### 7. Data Reporting / Regulatory Considerations

The SCa and NYS SEER research teams will independently contact participants, collect data and enter survey results in a unified study database maintained at USC. A Study ID will be created for each case and survey and registry data will be linked to it, and no personal identifiers (or registry IDs) will be included in the analytic dataset. Only staff directly involved with the study at each site will have access to the tracking systems. In addition, a central database will be maintained at Weill Cornell to assess the overall progress of the project. Each site will maintain a local password-protected and secure linkage database containing participant protected health information and identifiers and the linkage to the Study ID number. This database will only be accessible to researchers at the local site where the participant is followed. Participants will return their questionnaires to the local investigators. Accordingly, local study staff will go over each completed questionnaire and check all coding (although the questionnaire will be designed to be self-coded when possible).

#### 7.1 Institutional Review Board/Ethics Committee Approval

As required by local regulations, the Investigator will ensure all legal aspects are covered, and approval of the appropriate regulatory bodies obtained, before study initiation.

Before initiation of the study at each study center, the protocol, the ICF, other written material given to the patients, and any other relevant study documentation will be submitted to the appropriate Ethics Committee. Written approval of the study and all relevant study information must be obtained before the study center can be initiated. Any necessary extensions or renewals of IEC/IRB approval must be obtained for changes to the study, such as amendments to the protocol, the ICF, or other study documentation. The written approval of the IEC/IRB together with the approved ICF must be filed in the study files.

The Investigator will report promptly to the IEC/IRB any new information that may adversely affect the safety of the subjects or the conduct of the study. The Investigator will submit written summaries of the study status to the IEC/IRB as required. On completion of the study, the IEC/IRB will be notified that the study has ended.

All agreed protocol amendments will be clearly recorded on a protocol amendment form and will be signed and dated by the original protocol approving signatories. All protocol amendments will be submitted to the relevant institutional IEC/IRB for approval before implementation, as required by local regulations. The only exception will be when the amendment is necessary to eliminate an immediate hazard to the trial participants. In this case, the necessary action will be taken first, with the relevant protocol amendment following shortly thereafter.

Once protocol amendments or consent form modifications are implemented at the lead site, Weill Cornell Medicine, updated documents will be provided to participating sites. Weill Cornell Medicine must approve all consent form changes prior to local IRB submission.

Relevant study documentation will be submitted to the regulatory authorities of the participating countries, according to local/national requirements, for review and approval before the beginning of the study. On completion of the study, the regulatory authorities will be notified that the study has ended.

#### 7.2. Ethical Conduct of the Study

The Investigators and all parties involved should conduct this study in adherence to the ethical principles based on the Declaration of Helsinki, GCP, ICH guidelines and the applicable national and local laws and regulatory requirements.

This study will be conducted under a protocol reviewed and approved by the applicable ethics committees and investigations will be undertaken by scientifically and medically qualified persons, where the benefits of the study are in proportion to the risks.

#### 7.3 Informed Consent

The investigator or qualified designee must obtain documented consent according to ICH-GCP and local regulations, as applicable, from each potential subject or each subject's legally authorized representative prior to participating in the research study. Subjects who agree to participate will sign the approved informed consent form and will be provided a copy of the signed document.

The initial ICF, any subsequent revised written ICF and any written information provided to the subject must approved by IRB prior to use. The ICF will adhere to IRB/IEC requirements,

applicable laws and regulations.

#### 7.4 Compliance with Trial Registration and Results Posting Requirements

Under the terms of the Food and Drug Administration Modernization Act (FDAMA) and the Food and Drug Administration Amendments Act (FDAAA), the Sponsor-Investigator of the trial is solely responsible for determining whether the trial and its results are subject to the requirements for submission to <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>. Information posted will allow subjects to identify potentially appropriate trials for their disease conditions and pursue participation by calling a central contact number for further information on appropriate trial locations and trial site contact information.

#### 7.5 Record Retention

Essential documents are those documents that individually and collectively permit evaluation of the study and quality of the data produced. After completion of the study, all documents and data relating to the study will be kept in an orderly manner by the Investigator in a secure study file. All subject medical records and other source documentation will be kept for the maximum time permitted by the hospital, institution, or medical practice.

#### 8. Statistical Considerations

The data structure for the patient reported outcomes is longitudinal, and data could be missing at certain time points (e.g. a patient provides data at 8 but not 12 months). We will use a general estimating equations approach using a Gaussian link-function and auto-regressive correlation. The covariates will adjust for adverse events (prostate cancer aggressiveness [low or intermediate risk], age [continuous], race [white, black, other], comorbidity score [Charlson Index]) plus baseline disease-specific HRQOL score; treatment group will be entered as four separate variables (e.g. PGA 1 or 0; RP 1 or 0; SBRT 1 or 0; IMRT 1 or 0) with AS as the reference group.

Because differences between groups will vary by time (e.g. large decreases in urinary function in the surgery group at month 8, smaller by month 12), we will include a time by treatment interaction term. This model provides adjusted differences from AS over time for each treatment, along with a 95% CI and a p-value. From these estimates, it is straightforward to conduct pairwise comparisons (e.g. sexual function between PGA and surgery). As a sensitivity analysis, we will use propensity scores as the covariate as described above, again excluding patients at the extremes of the propensity distribution.

Adverse events will be treated as binary variables, defined as present or absent, with the severity being characterized by the associated categorical response. Mild AEs (grade 1) will be excluded because it typically resolves without intervention. However, inclusion of mild AEs will be considered in sensitivity analysis. Type and severity of AEs will be described separately by treatment.

The analysis will be by binomial logistic regression. The covariates will be age (continuous), BMI (using restricted cubic splines with knots at 30 and 35), comorbidity score (Charlson index), clinical stage (T1c or T2a, T2b, T2c, T3/4), NCCN risk group and pretreatment PSA (CI-5). Treatment group will be entered as 3 separate variables (i.e. PGA 1 or 0; SBRT 1 or 0; IMRT 1 or 0) with surgery as the reference group.

We will also conduct a sensitivity analysis using propensity methods – where propensity for treatment is derived from a multinomial logistic regression with the same covariates as above – and excluding any patient with >95% or <15% chance of receiving any of the treatments.

For adverse events, we expect a rate of 10% in the IMRT and RP arms. The main HRQOL endpoint of interest is EPIC-26 sexual function. The estimated number of patients we will evaluate is as follows: AS 300; PGA: 280; SBRT: 288; IMRT: 316; RP: 333. This is based on the incidence of low and intermediate prostate cancer in the SCa and NYS SEER registries.

## APPENDIX A.

## **Baseline Survey**

- 2. What is your birth date: \_\_\_\_/\_\_\_/19\_\_\_\_
- 3. When were you first diagnosed with prostate cancer: \_\_\_\_\_\_/\_\_\_/20\_\_\_\_\_
- 4. In general, you would say your health is:
  - ☐ Excellent
  - ☐ Very good
  - ☐ Good
  - ☐ Fair
  - ☐ Poor
  - ☐ Very poor
- 5. What is your most recent PSA result? \_\_\_\_\_ Don't know
- 6. What date was this PSA test done? \_\_\_\_ / \_\_ / 2 0 \_\_\_ Don't know
- 7. This next question is about your plans for treatment for prostate cancer or treatment you have already received.

For each of the following types of treatment, please indicate if you have chosen it, started to receive it, are considering it, or are not considering it at this time. Check one box on each row that best reflects your decision at this time for each type of treatment.

| Type of Treatment | this plan and chosen this completed it chosen this complete chosen this c | | I am considering this option but have not made a decision yet | I am not<br>considering<br>this option<br>at this time |
|---|---|---|---|---|
| a. Active Surveillance (My doctor will monitor how I am doing without directly treating the cancer) | Date started: // MM D D Y Y | | | |
| Type of Treatment (Cont.) | I have chosen<br>this plan and<br>have started or | I have<br>chosen this<br>plan but | I am<br>considering<br>this option but | I am not considering this option |

| | | completed it | have not yet received it | have not made a decision yet |
|---|---|---|---|---|
| b. | Prostate surgery<br>(radical<br>prostatectomy), which<br>would remove the<br>whole prostate. | Date of surgery: ——/——/—— M M D D Y Y | | |
| C. | HIFU / High Intensity<br>Focused Ultrasound<br>(ultrasound waves<br>cross tissue to destroy<br>the part of the prostate<br>that had cancer) | Date started: ——/——/—— M M D D Y Y | | |
| d. | <b>Cryotherapy</b> (freezing the <b>part</b> of the prostate that had cancer) | Date started: ——/——/—— MM D D Y Y | | |
| e. | Laser therapy | Date started: ——/——/—— MM D D Y Y | | |
| f. | Radio Frequency<br>Ablation | Date started: ——'——'—— MM D D Y Y | | |
| g. | Photodynamic<br>therapy | Date started: ——/——/—— MM D D Y Y | | |
| h. | External Beam<br>Radiation Therapy or<br>IMRT (radiation<br>treatment requiring<br>more than 2 weeks of<br>treatment) | Date started: // MM D D Y Y | | |
| i. | Stereotactic Body<br>Radiation Therapy<br>(SBRT) (radiation<br>treatment requiring<br>less than 2 weeks of<br>treatment) | Date started: ——/——/—— MM D D Y Y | | |

| j. Brachytherapy<br>(radioactive seeds)<br>This involves having<br>radioactive seeds<br>placed within the<br>prostate | Date started: '' M M D D Y Y |
|---|---|
| k. Proton Beam<br>Therapy | Date started: MM D D Y Y |
| I. Any other type of radiation therapy? Describe: | Date started: / MM D D Y Y |
| m. Hormonal treatments<br>to lower testosterone<br>(e.g. Lupron, Zoladex,<br>Firmagon, Eligard,<br>Vantas, etc) | Date started: ——/——/—— MM D D Y Y |
| n. Surgical removal of<br>testicles<br>(Orchiectomy) | Date of surgery: ——/——/—— MM D D Y Y |
| o. Chemotherapy<br>(docetaxel,<br>cabazitaxel, other) | Date started: |

<u>Health Before Treatment</u>
For the next set of questions, please refer to the time <u>just BEFORE you were diagnosed</u>.

## **Urinary Issues**

8. **During the 4 weeks before your diagnosis**, how often have you leaked urine (pee)? (Choose one)

| _ | More than once a day About once a day | | | | | |
|---|---|---|---|---|---|---|
| $\Box$ | More than once a week | | | | | |
| $\overline{\Box}$ | About once a week | | | | | |
| | Rarely or never | | | | | |
| 9. | Which of the following best describes yo diagnosis? (Choose one) | our urinary con | trol (ability to h | old pee) <b>durin</b> | g the 4 weeks | before your |
| | No urinary control whatsoever | | | | | |
| | Frequent dribbling | | | | | |
| | Occasional dribbling | | | | | |
| | Total control | | | | | |
| 10. | . How many pads or adult diapers per da before your diagnosis? (Choose one) | | lly use to contr | ol leakage (pe | e) during the 4 | weeks |
| | None | | | | | |
| | 1 pad per day | | | | | |
| | 2 pads per day | | | | | |
| | 3 or more pads per day | | | | | |
| | . How big a problem, if any, has each of (Choose one for each item) | the following be | een for you <b>du</b> i | ring the 4 wee | ks before you | diagnosis? |
| | | No<br>problem | Very<br>small<br>problem | Small<br>problem | Moderate<br>problem | Big<br>problem |
| a. | Dripping or leaking urine (pee) | | | | | |
| b. | Pain or burning on urination (when peeing) | | | | | |
| C. | Bleeding with urination (pee) | | | | | |
| d. | Weak urine stream (pee) or incomplete emptying | | | | | |
| e. | Need to urinate (pee) frequently during the day | | | | | |
| 12. | . Overall, how big a problem has your uri<br>your diagnosis? (Choose one) | nary function (a | ability to pee) b | peen for you <b>du</b> | ıring the 4 wee | ks before |
| П | No problem | | | | | |
| | Very small problem | | | | | |
| | Small problem | | | | | |
| | Moderate problem | | | | | |

| | Big problem | | | | | |
|---|---|---|---|---|---|---|
| 13. | Bowel Issues 13. How big a problem, if any, has each of the following been for you during the 4 weeks before your diagnosis? (Choose one response on each line) | | | | | |
| | | No<br>problem | Very<br>small<br>problem | Small<br>problem | Moderate<br>problem | Big<br>problem |
| a. | Urgency to have a bowel movement (poop) | | | | | |
| b. | Increased frequency of bowel movements (poop) | | | | | |
| C. | Losing control of your stools (poop) | | | | | |
| d. | Bloody stools (blood with poop) | | | | | |
| e. | Abdominal/pelvic/rectal pain | | | | | |
| | Overall, how big a problem have your byour diagnosis? (Choose one) | powel habits (ab | ility to poop) b | een for you <b>d</b> u | iring the 4 wee | ks before |
| | No problem<br>Very small problem<br>Small problem<br>Moderate problem<br>Big problem | | | | | |
| Sex | ual Issues | | | | | |
| | How would you rate each of the followi | ng <b>during the 4</b> | weeks before | e your diagno | sis? | |
| | Choose one response on each line) | Very poor to none | Poor | Fair | Good | Very<br>good |
| a. | Your ability to have an erection (hard on)? | | | | | |
| b. | Your ability to reach orgasm (climax)? | | | | | |
| | How would you describe the usual QU. diagnosis? (Choose one) | ALITY of your e | rections (hard | on) <b>during the</b> | e 4 weeks befo | re your |
| □ 1 | None at all | | | | | |
| | Not firm enough for any sexual a | activity | | | | |

| | Firm enough for masturbation an<br>Firm enough for intercourse | d foreplay o | nly | | | |
|---|---|---|---|---|---|---|
| 17. | 7. How would you describe the FREQUENCY of your erections (hard on) during the 4 weeks before your diagnosis? (Choose one) | | | | | |
| | I NEVER had an erection when I had an erection LESS THAN HAD I had an erection ABOUT HALF I had an erection MORE THAN HI had an erection WHENEVER I | ALF the time<br>the time I wa<br>HALF the tim | e I wanted or<br>anted one | | | |
| 18. | Overall, how would you rate your ability (Choose one) | to function sex | kually <b>during tl</b> | ne 4 weeks be | efore your diag | nosis? |
| | Very poor<br>Poor<br>Fair<br>Good<br>Very good | | | | | |
| | Overall, how big a problem has your set before your diagnosis? (Choose one) No problem Very small problem Small problem Moderate problem Big problem How big a problem during the 4 weeks response on each line) | | | | | |
| | | No<br>problem | Very<br>small<br>problem | Small<br>problem | Moderate<br>problem | Big<br>problem |
| a. | Feeling depressed | | | | | |
| b. | Lack of energy | | | | | |
| C. | Change in body weight | | | | | |
| _ | mographic Questions What is your ethnicity? Hispanic or Latino Not Hispanic or Latino | | | | | |

22. What is your race? (Choose all that apply)

| | White or Caucasian Black or African-American Asian Native Hawaiian or Other Pacific Islander Native American or Alaska Native |
|---|---|
| 23. | sat is your current marital status? Single or never married Married or domestic partnership Divorced Widowed Separated |
| 24. | at is your current employment status? Working full time Working part time Retired Unemployed or looking for work On disability |
| 25. | at is the HIGHEST level of education you have completed? Grade school or less Some high school High school graduate or GED Vocational school Some college Associates degree College graduate (Bachelor's degree) Some graduate education Graduate degree |
| 26. | <br>at is the total income of your household? Less than \$10,000 \$10,001 to \$20,000 \$20,001 to \$40,000 \$40,001 to \$70,000 \$70,001 to \$90,000 More than \$90,000 |

| | Private insurance (please select type below): |
|---|---|
| | ☐ Insurance provided through my current or former employer or union (including Kaiser/HMO/PPO) |
| | ☐ Insurance provided by another family member (e.g., spouse) through their current or former employer or union (including Kaiser/HMO/PPO) |
| | ☐ Insurance purchased directly from an insurance company (by you or another family member) |
| | ☐ Insurance purchased from an exchange (sometimes called Obamacare or the Affordable Care Act) |
| | Public or government insurance (please select type below): |
| | ☐ Medicaid or other state provided insurance |
| | ☐ Medicare/government insurance for age 65 years and older |
| | ☐ Medicare Advantage |
| | ☐ MediGAP |
| | VA (including those who have ever used or enrolled for VA health care) |
| П | I do not have any medical insurance |

# First Follow Up Survey

| 1. | Today's date: $\frac{1}{M} \frac{1}{M} \frac{1}{D} \frac{1}{D} \frac{1}{Y} \frac{1}{Y}$ | |
|---|---|---|
| 2. | How tall are you? (feet, inches) | |
| 3. | What is your weight?(pounds) | |
| 4. | Do you have any history of any of the following (check box | if Yes)?: |
| | ☐ Heart attack ☐ Congestive heart failure | Liver disease: Mild liver disease Moderate or severe liver disease |
| | □ Peripheral vascular disease | <u>Diabetes</u> : Diabetes without chronic complications Diabetes with chronic complications |
| | ☐ Cerebrovascular disease | |
| | ☐ Hypertension | |
| | ☐ Chronic pulmonary disease | ☐ Hemiplegia or paraplegia |
| | □ Rheumatologic disease | □ Renal disease |
| | □ Peptic ulcer disease | ☐ Any other malignancy besides prostate cancer, including leukemia and lymphoma |
| | | ☐ Metastatic (non-prostate) solid tumor |
| 5. | What was your last PSA value? (approximate value): | ng/ml |
| 6. | When was the date of your last PSA? (approximate date): | |
| | | Month Year |
| | | ☐ Don't know |

Choose one response on each line Not A little Quite Very Somewhat at all bit a bit much a. I keep close track of my PSA b. Knowing my PSA level is comforting to me П П П П c. I live in fear that my PSA will rise  $\square$ 8. Since your initial treatment for prostate cancer, did your doctor ever tell you that your prostate cancer came back (recurred) or progressed (got worse)? ☐ Yes □ No 9. Since you were diagnosed with prostate cancer, has a doctor ever told you that your prostate cancer had spread to other areas of your body? ☐ Yes □ No 10. These next guestions are about the treatments for prostate cancer that you have received. For each of the following types of treatment, please check the one(s) you have received and indicate the date you received it (or started it) I have received this Date received or **Type of Treatment** treatment started П a. Active Surveillance (My doctor will monitor how /\_\_\_/ I am doing without directly treating the cancer) D D Y Y ΜМ Prostate surgery (radical prostatectomy), which would remove the whole prostate. D D ΥY c. HIFU / High Intensity Focused Ultrasound (ultrasound waves cross tissue to destroy the ΜМ D D Y Y part of the prostate that had cancer) d. Cryotherapy (freezing the part of the prostate that had cancer) MM DD YY e. Laser therapy D D ΥΥ ММ

7. PSA: How true has each of the following statements been for you during the past 4 weeks?

f. Radio Frequency Ablation

D D

ΥY

ΜМ

| Type of | Treatment | I have received this treatment | Date received or started |
|---|---|---|---|
| g. | Photodynamic therapy | | //<br>MM D D Y Y |
| h. | External Beam Radiation Therapy or IMRT (radiation treatment requiring more than 2 weeks of treatment) | | //<br>MM D D Y Y |
| i. | Stereotactic Body Radiation Therapy (SBRT) (radiation treatment requiring less than 2 weeks of treatment) | | //<br>MM D D Y Y |
| j. | Brachytherapy (radioactive seeds) This involves having radioactive seeds placed within the prostate | | //<br>MM D D Y Y |
| k. | Proton Beam Therapy | | //<br>MM D D Y Y |
| l. | Any other type of radiation therapy? | | // |
| Describ | ə: <u> </u> | | MM D Y Y |
| m. | Hormonal treatments to lower testosterone<br>(e.g. Lupron, Zoladex, Firmagon, Eligard,<br>Vantas, etc) | | //<br>MM D D Y Y |
| n. | Surgical removal of testicles (Orchiectomy) | | //<br>MM D D Y Y |
| О. | Chemotherapy (docetaxel, cabazitaxel, other) | | //<br>MM D D Y Y |

If you have only received active surveillance or have not had any treatment yet for your prostate cancer, please skip to Question 16.

11. As individuals go through treatment for cancer, they sometimes experience different symptoms and side effects. For each symptom below, please select the one response that best describes your experiences in the 7 days after your initial treatment choice (surgery, radiation, partial gland ablation).

| 1) Symptom: Al | odominal pain | | | |
|---|---|---|---|---|
| a. In the 7 days after your initial treatment, how often did you have pain in the abdomen (belly area)? | | | | |
| □<br>Never | □<br>Rarely | □<br>Occasionally | □<br>Frequently | ☐<br>Almost constantly |
| b. In the 7 days after your initial treatment, what was the <b>severity</b> of your <b>pain in the abdomen (belly area)</b> at its <b>worst</b> ? | | | | |
| □<br>None | □<br>Mild | □<br>Moderate | □<br>Severe | □<br>Very severe |

| c. In the 7 days after your initial treatment, how much did <b>pain in the abdomen (belly area) interfere</b> with your usual or daily activities? | | | | |
|---|---|---|---|---|
| □<br>Not at all | □<br>A little bit | □<br>Somewhat | □<br>Quite a bit | □<br>Very much |
| 2) Symptom: S | walling | | | |
| | a. In the 7 days after your initial treatment, how often did you have arm or leg swelling? | | | |
| □<br>Never | □<br>Rarely | □<br>Occasionally | □<br>Frequently | ☐<br>Almost constantly |
| b. In the 7 days after y | our initial treatment, wh | nat was the <b>severity</b> of y | our <b>arm or leg swelli</b> i | ng at its worst? |
| □<br>None | □<br>Mild | □<br>Moderate | □<br>Severe | □<br>Very severe |
| c. In the 7 days after y activities? | our initial treatment, ho | w much did arm or leg s | swelling interfere with | n your usual or daily |
| □<br>Not at all | ☐<br>A little bit | □<br>Somewhat | □<br>Quite a bit | □<br>Very much |
| 3) Symptom: G | Seneral pain | | | |
| a. In the 7 days after y | our initial treatment, ho | ow <b>often</b> did you have <b>pa</b> | in? | |
| □<br>Never | □<br>Rarely | □<br>Occasionally | □<br>Frequently | ☐<br>Almost constantly |
| b. In the 7 days after y | our initial treatment, wh | nat was the <b>severity</b> of y | our <b>pain</b> at its worst? | |
| □<br>None | □<br>Mild | □<br>Moderate | □<br>Severe | □<br>Very severe |
| c. In the 7 days after y | our initial treatment, ho | w much did pain interfe | re with your usual or o | laily activities? |
| □<br>Not at all | □<br>A little bit | □<br>Somewhat | □<br>Quite a bit | □<br>Very much |
| 4) Symptom: F | atique | | | |
| | | nat was the <b>severity</b> of y | our <b>fatigue, tiredness</b> | s, or lack of energy at |
| □<br>None | □<br>Mild | □<br>Moderate | □<br>Severe | □<br>Very severe |
| b. In the 7 days after y your usual or daily act | | ow much did fatigue, tire | dness, or lack of ene | ergy interfere with |
| □<br>Not at all | □<br>A little bit | □<br>Somewhat | □<br>Quite a bit | □<br>Very much |

| 12. | Have you been hospitalized for complications from your prostate cancer treatment or for any other problems after receiving prostate cancer treatment? ☐ Yes: |
|---|---|
| | a. What was the reason for the hospitalization? |
| | b. How many days did you spend in the hospital? |
| | □ No |
| 13. | Did you perform Kegel exercises after your prostate cancer treatment? ☐ YesHow often do you (did you) do Kegel exercises? ☐ Once a week or less ☐ Twice a week ☐ More often than twice a week ☐ No ☐ I don't know |
| 14. | Did your doctor advise you to do Kegel exercises after your prostate cancer treatment? ☐ YesWhat resources were given to you to help you do Kegel exercises? Check all that apply. ☐ Verbal explanation ☐ Handout ☐ Visit with a Nurse Counselor ☐ Referral to Physical Therapy ☐ None ☐ I don't know ☐ Other: |
| | □ No □ I don't know |
| 15. | Did you experience any (other) complication or unexpected outcome within 3 months after your prostate cancer treatment? |
| | ☐ Yes: If yes, please describe: |
| | □ No |
| <u>Cur</u> | rent Health |
| 16. | In general, would you say your health is: |
| | □ Excellent □ Very good □ Good □ Fair □ Poor □ Very poor |
| Urir | the next set of questions, please think about your experience during the past 4 weeks. In the past 4 weeks how often did you leak urine (pee)? (Choose one) |
| □ M<br>□ A<br>□ M | flore than once a day bout once a day flore than once a week bout once a week arely or never |

| | Nhich of the following best describes y (Choose one) | our urinary con | trol (ability to h | old pee) <b>durin</b> | g the past 4 w | eeks? |
|---|---|---|---|---|---|---|
| | o urinary control whatsoever<br>equent dribbling<br>ccasional dribbling<br>tal control | | | | | |
| | How many pads or adult diapers did yo weeks? (Choose one) | u usually use p | er day to contro | ol urine (pee) l | eakage <b>during</b> | the past 4 |
| □ 2 p | one<br>oad per day<br>oads per day<br>or more pads per day | | | | | |
| 20. H | How big a problem, if any, was each of | the following d | uring the past | 4 weeks? (C | hoose one for e | ach item) |
| | | No problem | Very small problem | Small problem | Moderate problem | Big<br>problem |
| a. | Dripping or leaking urine (pee) | | | | | |
| b. | Pain or burning on urination (when peeing) | | | | | |
| C. | Bleeding with urination (when peeing) | | | | | |
| d. | Weak urine stream (pee) or incomplete emptying | | | | | |
| e. | Need to urinate (pee) frequently during the day | | | | | |
| C | Overall, how big a problem was your ur | rinary function ( | ability to pee) for | or you <b>during</b> | the past 4 wee | eks? (Choose |
| □ Ve<br>□ Sn<br>□ Mo | o problem<br>ery small problem<br>nall problem<br>oderate problem<br>g problem | | | | | |
| 22. ł | el Issues<br>How big a problem, if any, was each of<br><i>ine</i> ) | the following <b>d</b> | uring the past | 4 weeks? (C | hoose one resp | onse on each |
| | | No problem | Very small problem | Small problem | Moderate problem | Big<br>problem |
| a. | Urgency to have a bowel movement (poop) | | | | | |
| b. | Increased frequency of bowel movements (poop) | | | | | |
| C. | Losing control of your stools (poop) | | | | | |
| d. | Bloody stools (blood with poop) | | | | | |
| 0 | Abdominal/pelvic/rectal pain | П | П | П | П | П |

| 23. | Overall, how big a problem were your b | oowel habits (abi | lity to poop) d | uring the pas | t 4 weeks? (C | choose one) |
|---|---|---|---|---|---|---|
| □ Ve<br>□ Sr<br>□ M | o problem<br>ery small problem<br>mall problem<br>oderate problem<br>g problem | | | | | |
| 24. | ual Issues Do you currently use any of the followine each line) | ng to help with p | roblems with s | sexual function | ? (Choose one | e response on |
| | | | | | Yes | No |
| a. | Vacuum suction device | | | | | |
| b. | Penile injections (shots) | | | | | |
| C. | Pills, such as Viagra, Cialis, Levitra, | Staxyn, Stendra | | | | |
| d. | Urethral pellets or suppositories (Mu | se) | | | | |
| e. | Penile prosthesis (surgical implant) | | | | | |
| f. | Other (please specify): | | | | | |
| 25. | How would you rate each of the followi (Choose one response on each line) | ng <b>during the p</b> Very poor | | Fair | Cood | Vorugoed |
| | | to none | Poor | rair | Good | Very good |
| a. | Your ability to have an erection (getting hard for sex)? | | | | | |
| b. | Your ability to reach orgasm (climax)? | | | | | |
| | How would you describe the usual QU<br>(Choose one) | ALITY of your er | ections (gettin | g hard for sex | ) during the p | ast 4 weeks? |
| □ No | one at all<br>ot firm enough for any sexual activity<br>rm enough for masturbation and forepl<br>rm enough for intercourse | ay only | | | | |
| | How would you describe the FREQUE (Choose one) | NCY of your ered | ctions (getting | hard for sex) | during the pa | st 4 weeks? |
| <br> <br> | NEVER had an erection when I wanted had an erection LESS THAN HALF the had an erection ABOUT HALF the time had an erection MORE THAN HALF the had an erection WHENEVER I wanted | time I wanted or<br>I wanted one<br>e time I wanted o | | | | |
| 28. | Overall, how would you rate your ability | y to function sex | ually <b>during tl</b> | ne past 4 wee | ks? (Choose | one) |
| □ Po<br>□ Fa<br>□ Go | air | | | | | |

| V No □ No □ Ve □ Sm □ Mo | Overall, how big a problem was your veeks? (Choose one) problem ry small problem hall problem derate problem g problem How often have you been able to eja | | | | you <b>during the</b> | past 4 |
|---|---|---|---|---|---|---|
| ☐ Mo<br>☐ Ab<br>☐ Le: | the time set of the time out half the time se than half the time ne of the time / could not ejaculate | | | | | |
| 31. F | How would you rate the strength or f | orce of your ejacu | ulation? | | | |
| ☐ A I<br>☐ So<br>☐ Mu<br>☐ Ve | □ As strong as it always was □ A little less strong than it used to be □ Somewhat less strong than it used to be □ Much less strong than it used to be □ Very much less strong than it used to be □ Could not ejaculate | | | | | |
| 32. F | low would you rate the amount or v | olume of semen of | or fluid when yo | u ejaculate? | | |
| □ A I<br>□ So<br>□ Mu<br>□ Ve | much as it always was ittle less than it used to be mewhat less than it used to be ich less than it used to be ry much less than it used to be uld not ejaculate | | | | | |
| 33. I | f you have had any ejaculation diffic | ulties or have bee | en unable to eja | iculate, have y | ou been bother | ed by this? |
| □ No □ A I □ Mo □ Ve | □ No problem with ejaculation □ Not at all bothered □ A little bothered □ Moderately bothered □ Very bothered □ Extremely bothered | | | | | |
| | How big a problem <b>during the past</b> <i>ine)</i> | <b>4 weeks</b> was eac | ch of the following | ng for you? (C | hoose one resp | onse on each |
| | | No problem | Very small problem | Small<br>problem | Moderate problem | Big<br>problem |
| a. | Feeling depressed | | | | | |
| b. | Lack of energy | | | | | |
| C. | Change in body weight | | | | | |

The best health For the next set of questions, indicate which best describes your health TODAY. you can imagine 35. Mark an **X** on the scale to indicate how your health is **today**. 100 This scale is numbered from 0 to 100. 100 means the best health you can imagine. 95 0 means the worst health you can imagine. 90 85 Please write the number you marked on the scale in the box: 36. Mobility: 80 ☐ I have no problems walking □ I have slight problems walking 75 ☐ I have moderate problems walking ☐ I have severe problems walking 70 ☐ I am unable to walk 37. Self-care: 65 ☐ I have no problems washing or dressing myself ☐ I have slight problems washing or dressing myself 60 ☐ I have moderate problems washing or dressing myself ☐ I have severe problems washing or dressing myself 55 ☐ I am unable to wash or dress myself 38. Usual activities 50 (e.g. work, study, housework, family or leisure activities): ☐ I have no problems doing my usual activities 45 ☐ I have slight problems doing my usual activities ☐ I have moderate problems doing my usual activities 40 ☐ I have severe problems doing my usual activities ☐ I am unable to do my usual activities 35 39. Pain / Discomfort: ☐ I have no pain or discomfort 30 ☐ I have slight pain or discomfort ☐ I have moderate pain or discomfort ☐ I have severe pain or discomfort 25 ☐ I have extreme pain or discomfort 40. Anxiety / Depression 20  $\hfill\square$  I am not anxious or depressed ☐ I am slightly anxious or depressed 15 ☐ I am moderately anxious or depressed ☐ I am severely anxious or depressed ☐ I am extremely anxious or depressed 10 5 0 The worst health you can imagine

## Views Surrounding Impact of Prostate Cancer and Treatment Decision

| 41. | During the past four weeks, how much of the tkind of treatment you chose for your prostate call All of the time ☐ Most of the time ☐ A good bit of the time ☐ Some of the time ☐ A little bit of the time ☐ None of the time | • | shed that you o | could change you | ir mind about the |
|---|---|---|---|---|---|
| 42. | <ul> <li>2. How true or false has the following statement been for you during the past four weeks: <ul> <li>I feel that I would be better off if I had chosen the other treatment for prostate cancer.</li> <li>Definitely true</li> <li>Mostly true</li> <li>Neither true nor false</li> <li>Mostly false</li> <li>Definitely false</li> </ul> </li> </ul> | | | | |
| 43. | How true or false has the following statement be It bothers me that other men with prostate cance Definitely true Mostly true Neither true nor false Mostly false Definitely false | | | | have received. |
| 44. | Listed below are a number of statements concer week, please indicate how much you agree or d | isagree with each | | ieir own health. <b>C</b> | |
| | | Strongly agree | Agree | Disagree | Strongly<br>Disagree |
| a. | Because cancer is unpredictable, I feel I cannot plan for the future. | | | | |
| b. | My fear of having my cancer getting worse gets in the way of enjoying life. | | | | |
| C. | I am afraid of my cancer getting worse. | | | | |
| d. | I am more nervous since I was diagnosed with prostate cancer. | | | | |

| 45. | 5. Outlook: How true is each of the following statements for you? (Choose one response on each line) | | | | | |
|---|---|---|---|---|---|---|
| | | Not at all | A little bit | Somewhat | Quite a bit | Very much |
| a. | I feel that my cancer has given me a better outlook on life. | | | | | |
| b. | I feel that coping with cancer has made me a stronger person. | | | | | |
| 46. | Are there any other issues or concerns mention? | about your pro | state cancer o | r your treatmen | t that you woul | d like to |

Thank you very much for completing this survey. Please return in one of the enclosed postage paid envelopes or mail to address on front of survey.

Please also review and complete the HIPAA form if you agree to provide authorization for us to review your medical records regarding your prostate cancer and treatment.

# Second Follow Up Survey

## **General Questions**

| 1. | Today's date://20 | _ | | | | |
|---|---|---|---|---|---|---|
| | M M D D Y Y | / Y Y | | | | |
| 2. | What was your last PSA value? (approximate | e value): | · <u>-</u> | ng/ml | | |
| | | | | Don't know | | |
| 3. | When was the date of your last PSA? (appro | ximate da | ite):/_ | | | |
| | | | Month | Year | | |
| | | | | Don't know | | |
| 4. | PSA: How true has each of the following sta<br>Choose one response on each line. | tements b | een for you duri | ing the <b>past 4 we</b> | eks? | |
| | | Not<br>at all | A little<br>bit | Somewhat | Quite<br>a bit | Very<br>much |
| a. | I keep close track of my PSA | | | | | |
| b. | Knowing my PSA level is comforting to me | | | | | |
| C. | I live in fear that my PSA will rise | | | | | |
| 5. | Since your initial treatment for prostate cance (recurred) or progressed (got worse)? ☐ Yes ☐ No | er, did you | ur doctor ever te | ll you that your p | rostate cai | ncer came back |
| 6. | Since you were diagnosed with prostate can to other areas of your body? ☐ Yes ☐ No | cer, has a | doctor ever tolo | d you that your pr | ostate car | icer had spread |
| 7. | These next questions are about the treatmer time (even if you have told us about them For each of the following types of treatment, received it (or started it): | before). | | - | - | - |
| | Type of Treatment | _ | ve received this | s Date recei<br>started | ved or | |
| | Active Surveillance (My doctor will moniton how I am doing without directly treating the cancer) | | | / | _/<br>D YY | |
| | Prostate surgery (radical prostatectomy which would remove the whole prostate. | ), | | / | _/ | |

MM DD YY

| HIFU / High Intensity Focused Ultrasound<br>(ultrasound waves cross tissue to destroy the<br>part of the prostate that had cancer) | ///<br>MM D D Y Y |
|---|---|
| <b>Cryotherapy</b> (freezing the <b>part</b> of the prostate that had cancer) | / |
| Laser therapy | //<br>MM D D Y Y |
| Radio Frequency Ablation | //<br>MM D D Y Y |
| Photodynamic therapy | //<br>MM D D Y Y |
| External Beam Radiation Therapy or IMRT (radiation treatment requiring more than 2 weeks of treatment) | / |
| Stereotactic Body Radiation Therapy<br>(SBRT) (radiation treatment requiring less<br>than 2 weeks of treatment) | //<br>MM D D Y Y |
| Brachytherapy (radioactive seeds) This involves having radioactive seeds placed within the prostate | / |
| Proton Beam Therapy | //<br>MM D D Y Y |
| Any other type of radiation therapy? Describe: | //<br>MM D D Y Y |
| Hormonal treatments to lower<br>testosterone (e.g. Lupron, Zoladex,<br>Firmagon, Eligard, Vantas, etc) | //<br>MM D D Y Y |
| Surgical removal of testicles (Orchiectomy) | //<br>MM D D Y Y |
| Chemotherapy (docetaxel, cabazitaxel, other) | //<br>MM D D Y Y |

| How did you make your treatment decision? |
|---|
| ☐ I made the decision alone |
| ☐ I made the decision together with a family member or friend |
| ☐ I made the decision together with my doctor, nurse, or health practitioner |
| $\square$ I made the decision together with a family member or friend and my doctor, nurse, or health practitioner |
| ☐ My doctor, nurse, or health practitioner made the decision |
| ☐ I don't know or remember how the decision was made |

8.

| 9. | What were the most important factors you considered in making your treatment decision? (Check all that apply) Best chance for cure of my cancer Minimize side effects related to sexual function Minimize side effects related to urinary function |
|---|---|
| | ☐ Minimize side effects related to bowel function |
| | ☐ Minimize financial cost ☐ Amount of time and travel required to receive treatments |
| | ☐ Length of recovery time |
| | ☐ Amount of time away from work |
| | ☐ Burden on family members ☐ Reduction of worry and concern about cancer |
| | Line Reduction of worry and concern about cancel |
| 10. | Have you been hospitalized for complications from your prostate cancer treatment or for any other problems after receiving prostate cancer treatment? ☐ Yes |
| | a. What was the reason for the hospitalization? |
| | b. How many days did you spend in the hospital? □ No |
| 11. | Did you experience any (other) complication or unexpected outcome within 3 months after your prostate cancer treatment? |
| | ☐ Yes: If yes, please describe: |
| | □ No |
| Cur | rent Health |
| | In general, would you say your health is: |
| | □ Excellent |
| | □ Very good |
| | □ Good |
| | □ Fair |
| | □ Poor |
| | □ Very poor |

## For the next set of questions, indicate which best describes your health **TODAY**.

| 13. | Mobility: ☐ I have no problems walking ☐ I have slight problems walking | The best health | |
|---|---|---|---|
| | <ul> <li>□ I have moderate problems walking</li> <li>□ I have severe problems walking</li> <li>□ I am unable to walk</li> </ul> | # | 100 |
| | | # | 95 |
| 14. | Self-care: ☐ I have no problems washing or dressing myself | # | |
| | ☐ I have slight problems washing or dressing myself | | 90 |
| | $\square$ I have moderate problems washing or dressing myself | # | 0.5 |
| | ☐ I have severe problems washing or dressing myself | 主 | 85 |
| | ☐ I am unable to wash or dress myself | # | |
| 15. | Usual activities | = | 80 |
| | (e.g. work, study, housework, family or leisure activities): | + | 75 |
| | ☐ I have no problems doing my usual activities | 王 | 75 |
| | ☐ I have slight problems doing my usual activities | + | 70 |
| | ☐ I have moderate problems doing my usual activities ☐ I have severe problems doing my usual activities | = | 70 |
| | ☐ I am unable to do my usual activities | 主 | 65 |
| | | # | 03 |
| 16. | Pain / Discomfort: | <u></u> | 60 |
| | ☐ I have no pain or discomfort ☐ I have slight pain or discomfort | 主 | 00 |
| | ☐ I have moderate pain or discomfort | 丰 | 55 |
| | ☐ I have severe pain or discomfort | 主 | 00 |
| | ☐ I have extreme pain or discomfort | <del>-</del> | 50 |
| | | 圭 | |
| 17. | Anxiety / Depression | + | 45 |
| | ☐ I am not anxious or depressed | <b>王</b> | |
| | ☐ I am slightly anxious or depressed ☐ I am moderately anxious or depressed | | 40 |
| | ☐ I am severely anxious or depressed | Ξ. | |
| | ☐ I am extremely anxious or depressed | + | 35 |
| | | # | |
| | | <del>-</del> | 30 |
| 18. | Mark an <b>X</b> on the scale to indicate how your health is <b>today</b> . | 主 | |
| | This scale is numbered from 0 to 100. | <del>+</del> | 25 |
| | 100 means the <u>best</u> health you can imagine. | 圭 | |
| | 0 means the worst health you can imagine. | + | 20 |
| | | <b>=</b> | |
| | | 主 | 15 |
| | Please write the number you marked on the scale in the box. | # | 40 |
| | <u></u> | = | 10 |
| | | 主 | 5 |
| | | = | 3 |
| | | _= | 0 |
| | | The worst healt you can imagin | |

| Urina | he next set of questions, please thinary Issues n the past 4 weeks how often did you | - | • | | 4 weeks. | |
|---|---|---|---|---|---|---|
| □ Ab □ Mo | ore than once a day<br>out once a day<br>ore than once a week<br>out once a week<br>urely or never | | | | | |
| | Nhich of the following best describes y Choose one) | our urinary con | trol (ability to h | old pee) <b>durin</b> | g the past 4 w | eeks? |
| | o urinary control whatsoever<br>equent dribbling<br>ccasional dribbling<br>tal control | | | | | |
| | How many pads or adult diapers did yo | ou usually use p | er day to contr | ol urine (pee) l | eakage <b>during</b> | the past 4 |
| □ 2 p | one<br>bad per day<br>bads per day<br>or more pads per day | | | | | |
| 22. H | How big a problem, if any, was each of | f the following <b>d</b><br>No problem | uring the past<br>Very small<br>problem | t <b>4 weeks</b> ? <i>(Cl</i><br>Small<br>problem | hoose one for e<br>Moderate<br>problem | ach item)<br>Big<br>problem |
| a. | Dripping or leaking urine (pee) | | | | | |
| b. | Pain or burning on urination (when peeing) | | | | | |
| C. | Bleeding with urination (when peeing) | | | | | |
| d. | Weak urine stream (pee) or incomplete emptying | | | | | |
| e. | Need to urinate (pee) frequently during the day | | | | | |
| □ No □ Ve □ Sn □ Mo | Overall, how big a problem was your u<br>one)<br>o problem<br>ory small problem<br>nall problem<br>oderate problem<br>g problem | rinary function ( | ability to pee) f | or you <b>during</b> | the past 4 wee | eks? (Choose |
| 24. H | el Issues<br>How big a problem, if any, was each of<br>ine) | f the following <b>d</b> | uring the past | t <b>4 weeks</b> ? (Cl | hoose one resp | onse on eacl |
| | | No problem | Very small problem | Small<br>problem | Moderate problem | Big<br>problem |
| a. | Urgency to have a bowel movement (poop) | | | | | |
| b. | Increased frequency of bowel movements (poop) | | | | | |

| C. | Losing control of your stools (poop) | | | | | |
|---|---|---|---|---|---|---|
| d. | Bloody stools (blood with poop) | | | | | |
| e. | Abdominal/pelvic/rectal pain | | | | | |
| 25. | Overall, how big a problem were your b | owel habits (abi | ility to poop) <b>d</b> | uring the pas | t 4 weeks? (C | Choose one) |
| □ Ve<br>□ Si<br>□ M | o problem<br>ery small problem<br>mall problem<br>oderate problem<br>g problem | | | | | |
| Sexu | ual Issues | | | | | |
| | Do you currently use any of the followin each line) | g to help with p | roblems with s | sexual function | • | • |
| | | | | | Yes | No |
| a. | Vacuum suction device | | | | | |
| b. | Penile injections (shots) | | | | | |
| C. | Urethral pellets or suppositories (Mus | se) | | | | |
| d. | Penile prosthesis (surgical implant) | | | | | |
| e. | Other (please specify): | | | | | |
| | How would you rate each of the followir (Choose one response on each line) | ng <b>during the p</b> | ast 4 weeks? | | | |
| | | Very poor to none | Poor | Fair | Good | Very good |
| a. | Your ability to have an erection (getting hard for sex)? | | | | | |
| b. | Your ability to reach orgasm (climax)? | | | | | |
| □ No | How would you describe the usual QUA (Choose one) one at all of firm enough for any sexual activity rm enough for masturbation and foreplarm enough for intercourse | · | ections (gettin | g hard for sex | ) during the p | ast 4 weeks? |
| | How would you describe the FREQUEN (Choose one) | NCY of your ered | ctions (getting | hard for sex) | during the pa | st 4 weeks? |
| | NEVER had an erection when I wanted had an erection LESS THAN HALF the thad an erection ABOUT HALF the time had an erection MORE THAN HALF the had an erection WHENEVER I wanted contact the second se | time I wanted or<br>I wanted one<br>time I wanted c | | | | |

| <ul><li>□ Ve</li><li>□ Po</li><li>□ Fa</li><li>□ Go</li></ul> | ıir | lity to function sex | rually <b>during t</b> h | ne past 4 wee | k <b>s</b> ? (Choose or | ne) |
|---|---|---|---|---|---|---|
| □ No □ Ve □ Sr | Overall, how big a problem was your weeks? (Choose one) o problem ery small problem nall problem oderate problem g problem | sexual function, o | or lack of sexua | l function, for y | you <b>during the</b> | past 4 |
| ☐ All<br>☐ Me<br>☐ All<br>☐ Le | How often have you been able to eja<br>I the time<br>ost of the time<br>bout half the time<br>ess than half the time<br>one of the time / could not ejaculate | culate or "cum" wi | hen having sex | ual activity? | | |
| □ As □ A □ Sc □ Mc | How would you rate the strength or for strong as it always was little less strong than it used to be somewhat less strong than it used to be such less strong than it used to be ery much less strong than it used to be bould not ejaculate | e | lation? | | | |
| ☐ As<br>☐ A<br>☐ So<br>☐ Mi | How would you rate the amount or voor much as it always was little less than it used to be somewhat less than it used to be such less than it used to be erry much less than it used to be bould not ejaculate | olume of semen o | r fluid when you | u ejaculate? | | |
| 35. | f you have had any ejaculation diffic | ulties or have bee | n unable to eja | culate, have y | ou been bother | ed by this? |
| □ No □ A □ Mo □ Ve | o problem with ejaculation<br>of at all bothered<br>little bothered<br>oderately bothered<br>ery bothered<br>tremely bothered | | | | | |
| | How big a problem <b>during the past</b> <i>d</i> | <b>4 weeks</b> was eac | h of the followir | ng for you? (Ci | hoose one resp | onse on each |
| | | No problem | Very small problem | Small<br>problem | Moderate problem | Big<br>problem |
| a. | Feeling depressed | | | | | |
| b. | Lack of energy | | | | | |
| C | Change in body weight | П | П | П | П | П |

## Views Surrounding Impact of Prostate Cancer and Treatment Decision

| | During the past four weeks, how much of the time have kind of treatment you chose for your prostate cancer? ☐ All of the time ☐ Most of the time ☐ A good bit of the time ☐ Some of the time ☐ A little bit of the time ☐ None of the time | e you wished th | nat you coul | d change your mi | nd about the |
|---|---|---|---|---|---|
| | How true or false has the following statement been for your Ifeel that I would be better off if I had chosen the other to Definitely true ☐ Mostly true ☐ Neither true nor false ☐ Mostly false ☐ Definitely false | | | | |
| | How true or false has the following statement been for your lt bothers me that other men with prostate cancer get treed Definitely true Mostly true Neither true nor false Mostly false Definitely false | | | | e received. |
| <b>Belo</b> 40. | w is a list of comments made by men about prostate Please indicate how frequently these comments were true | | _ | | - |
| | item) | Not at all | Rarely | Sometimes | Often |
| a. | Any reference to prostate cancer brought up strong feelings in me. | | | | |
| b. | Even though it's a good idea, I found that getting a PSA test scared me. | | | | |
| C. | Whenever I heard about a friend or public figure with prostate cancer, I got more anxious about my having prostate cancer | | | | |
| d. | When I thought about having a PSA test, I got more anxious about my having prostate cancer. | | | | |
| e. | Other things kept making me think about prostate cancer. | | | | |
| f. | I felt kind of numb when I thought about prostate cancer. | | | | |
| g. | I thought about prostate cancer even though I didn't mean to. | | | | |

| h. | I had a lot of feelings about prostate cancer, but I didn't want to deal with them. | | | | |
|---|---|---|---|---|---|
| i. | I had more trouble falling asleep because I couldn't get thoughts of prostate cancer out of my mind. | | | | |
| j. | I was afraid that the results from my PSA test would show that my disease was getting worse. | | | | |
| k. | Just hearing the words "prostate cancer" scared me | . 🗆 | | | |
| 41. | Please indicate how frequently these situations have <b>E</b> | EVER been true | e for you. | | |
| | | Not at all | Rarely | Sometimes | Often |
| a. | I have been so anxious about my PSA test that I have thought about delaying it. | | | | |
| b. | I have been so worried about my PSA test result that I have thought about asking my doctor to repeat it. | at 🗆 | | | |
| C. | I have been so concerned about my PSA test result that I have thought about having the test repeated a another lab to make sure they were accurate. | | | | |
| 42. | Listed below are a number of statements concerning a week, please indicate how much you agree or disagree | e with each sta | efs about theil<br>atement. | r own health. <b>Dur</b> | |
| | | trongly<br>agree | Agree | Disagree | Strongly<br>Disagree |
| a. | Because cancer is unpredictable, I feel I cannot plan for the future. | | | | |
| b. | My fear of having my cancer getting worse gets in the way of enjoying life. | | | | |
| C. | I am afraid of my cancer getting worse. | | | | |
| d. | I am more nervous since I was diagnosed with prostate cancer. | | | | |